CLINICAL TRIAL: NCT06822595
Title: High-Load Blood Flow Restriction (BFR) Training May Decrease Anaerobic Fatigue in Distance Runners: A Randomized Controlled Trial
Brief Title: High-Load Blood Flow Restriction (BFR) Training May Decrease Anaerobic Fatigue in Distance Runners
Acronym: BFR-Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Tuğba Kocahan, associate professor, Gulhane Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SBU-GTF
Record Dates: First submitted 2025-02-02; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Anaerobic Performance
Keywords: Athlete; muscular; KAATSU; sports medicine; performance
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood flow restriction (BFR) Group (Experimental): BFR group followed an identical 8-week isokinetic training protocol twice weekly. The BFR group performed exercises with arterial occlusion pressure set to 80% of the measured occlusion pressure.
  Interventions: Device: Blood flow restriction (BFR) training; Device: Isokinetic training
- Control Group (Active Comparator): Control group followed an identical 8-week isokinetic training protocol twice weekly.
  Interventions: Device: Isokinetic training

INTERVENTIONS:
Device: Blood flow restriction (BFR) training — Both groups followed an identical 8-week isokinetic training protocol twice weekly. The BFR group performed exercises with arterial occlusion pressure set to 80% of the measured occlusion pressure.
  Other Names: Isokinetic training
  Arms: Blood flow restriction (BFR) Group
Device: Isokinetic training — Both groups followed an identical 8-week isokinetic training protocol twice weekly.

SUMMARY:
This study investigates the effects of high-load BFR training on anaerobic performance and fatigue resistance in distance runners. To determine whether adding BFR to isokinetic resistance training improves anaerobic performance and 5-10 km running times in runners. Forty-two runners were randomized into BFR (n=21) and control (n=21) groups. Both groups followed an identical 8-week isokinetic training protocol twice weekly. The BFR group performed exercises with arterial occlusion pressure set to 80% of the measured occlusion pressure. Anaerobic performance was assessed via the Wingate test, and 5 km and 10 km running times were recorded before and after the intervention. Statistical analyses compared pre- and post-training performance within and between groups.

DETAILED DESCRIPTION:
Blood flow restriction (BFR) training is increasingly used to enhance athletic performance, but its effects on anaerobic fatigue in distance runners remain unclear. This study investigates the effects of high-load BFR training on anaerobic performance and fatigue resistance in distance runners.To determine whether adding BFR to isokinetic resistance training improves anaerobic performance and 5-10 km running times in runners.

Forty-two runners were randomized into BFR (n=21) and control (n=21) groups. Both groups followed an identical 8-week isokinetic training protocol twice weekly. The BFR group performed exercises with arterial occlusion pressure set to 80% of the measured occlusion pressure. Anaerobic performance was assessed via the Wingate test, and 5 km and 10 km running times were recorded before and after the intervention. Statistical analyses compared pre- and post-training performance within and between groups.

ELIGIBILITY:
Inclusion Criteria:

* The absence of cardiovascular or musculoskeletal conditions,
* No recent resistance training,
* Running more than 20 kilometers per week.

Exclusion Criteria:

* Having a cardiovascular or musculoskeletal condition,
* Having done recent resistance training,
* Running less than 20 kilometers per week.

Ages: 22 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
The effects of an isokinetic training program combined with blood flow restriction (BFR) on anaerobic performance and fatigue resistance in long-distance runners were investigated. | baseline and week 8
  Lower extremity Wingate Test (WanT) was used to evaluate the anaerobic capacities of long-distance runners. In calculating the fatigue index; (peak power - minimum power/peak power) x 100 (% fatigue index) formula was used.

CONTACTS AND LOCATIONS:
Overall Officials: Hüseyin Günaydın, Study Chair — University of Health Sciences, Gulhane Faculty of Medicine, Ankara/Türkiye
Locations (2):
- Turkey (Türkiye) (2):
  - Hüseyin Günaydın, Ankara
  - University of Health Sciences, Gulhane Faculty of Medicine, Ankara